CLINICAL TRIAL: NCT03835377
Title: A Randomized Feeding Trial of Iron-Biofortified Beans in School Children in Mexico
Brief Title: Iron-Biofortified Beans Intervention in Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CI-441
Record Dates: First submitted 2019-01-11; First posted 2019-02-08 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Iron-deficiency; Anemia
Keywords: Iron; Biofortification; Iron deficiency; Anemia; Children; Mexico
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study was a double-blind, cluster-randomized controlled trial (with randomization at the school level) of: (1) iron-biofortified black beans, compared to (2) a commercial variety of beans, with the intervention randomized at the school level. School administrators, children, research staff (i.e. managing the intervention, food weighing, assessment of outcomes), and laboratory staff were blinded to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron-biofortified beans (Experimental): Iron-biofortified beans (Phaseolus vulgaris L MIB465)
  Interventions: Other: Iron-biofortified beans
- Control beans (Active Comparator): Control beans (Phaseolus vulgaris L Jamapa variety)
  Interventions: Other: Control beans

INTERVENTIONS:
Other: Iron-biofortified beans — Iron-biofortified beans (Phaseolus vulgaris L MIB465)
  Other Names: Fe-Beans
  Arms: Iron-biofortified beans
Other: Control beans — Control beans (Phaseolus vulgaris L Jamapa variety), identical in color and size
  Other Names: Control-Beans
  Arms: Control beans

SUMMARY:
The objective of this cluster-randomized efficacy feeding trial was to determine the effects of consuming iron-biofortified beans (Fe-Beans) on iron status in children, compared to control beans (Control-Beans). A cluster-randomized trial of biofortified beans (Phaseolus vulgaris L), bred to enhance iron content, was conducted for 6 months.

DETAILED DESCRIPTION:
Iron deficiency is the most common single nutrient deficiency worldwide, with the highest burden in children and women of reproductive age. Global estimates of anemia prevalence in school-aged children range between 25% and 46%, and iron deficiency accounts for a majority of anemia cases. In Mexico, the national nutrition and health survey (2006) reported a prevalence of anemia of 16.6% and iron deficiency of 17.6% (serum ferritin <12.0 µg/L), posing a considerable health risk for children.

Interventions, including micronutrient supplementation and food fortification, have improved iron status and reduced the prevalence of anemia in some settings. However, iron deficiency remains an urgent public health problem and threat to child health and development. Young children are particularly at high risk due to rapid growth, inadequate dietary intake, and high risk of infection in resource-limited settings. Iron deficiency has been associated with impaired cognitive function in children, and long-term impairments in physical work capacity into adulthood.

One novel approach to reducing micronutrient malnutrition is to enhance the nutrient quality of the diet through biofortification of staple crops that are already locally accepted and consumed. Biofortification has consequently been recognized by the Copenhagen Consensus of 2008 as one of the top five solutions to current global health and nutrition challenges. The success and challenges of biofortification have been documented previously. We recently reviewed the published evidence from the three randomized efficacy trials of different iron-biofortified crops that demonstrated varied benefits in populations, including rice in adult Filipino women, pearl millet in school-aged children in India, and beans in women of reproductive age in Rwanda. Findings demonstrated improvements in serum ferritin concentrations and total body iron concentrations, with additional potential to benefit in individuals who were iron deficient at baseline. Given this limited evidence and with no studies from Latin America, more studies with diverse populations and locally relevant crops are warranted before implementation of a potentially important public health intervention.

In order to target at-risk populations in Latin America, the Centro Internacional de Agricultura Tropical (CIAT) in Colombia bred and biofortified a common black bean variety (Phaseolus vulgaris L), the standard black bean currently consumed widely in Central America and Mexico. In Mexico, beans have been ranked highly among the most consumed foods by school-aged children nationwide, according to Encuesta Nacional de Salud y Nutrición, a nationally representative nutrition survey in 2006. Biofortification has nearly doubled the iron concentration (~100 versus ~50 mg/kg) of the standard bean variety. We hypothesized that daily consumption of iron-biofortified beans (Fe-Beans) would improve hemoglobin, serum ferritin, and total body iron in 6 months, compared to control beans (Control-Beans). In order to examine this hypothesis, we conducted the first randomized efficacy trial of iron-biofortified beans and iron status in primary school-aged children in a low-income setting in Mexico. Special consideration was applied to assess indicators of iron status with and without anemia and measured inflammatory markers, which can mask iron deficiency, particularly in similar settings where the prevalence of infection is high.

The objective of this cluster-randomized efficacy feeding trial was to determine the effects of consuming iron-biofortified beans (Fe-Beans) on iron status in children, compared to control beans (Control-Beans).

The long-term goal of this study is to determine if iron bio-fortification of beans is an efficacious and potentially effective strategy to improve iron status of at-risk populations in resource-limited settings.

ELIGIBILITY:
Inclusion criteria:

* Boarding schools for children (5-12 y)
* Located in a rural area approximately 60 kilometers east of the city of Oaxaca
* A high prevalence of anemia (>=15.0%) on the baseline survey
* Adequate infrastructure to sustain a 6-month feeding trial. Exclusion criteria were a prevalence of anemia of less than 15% on the baseline survey, and inadequate infrastructure to sustain a 6-month feeding trial

Exclusion Criteria:

* A prevalence of anemia <15.0% on the baseline survey
* Inadequate infrastructure to sustain a 6-month feeding trial

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 574 (Actual)
Dates: Start 2010-01-06 (Actual); Primary Completion 2010-06-25 (Actual); Study Completion 2010-08-15 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin | 6 months
  Hemoglobin (Hb)
Change in serum ferritin | 6 months
  Serum ferritin (SF)
Change in sTfR | 6 months
  Soluble transferrin receptor (sTfR)
Anemia | 6 months
  Hb <115 g/L for <12 y; <120 g/L for >=12 y
Iron deficiency (SF) | 6 months
  Serum ferritin <15.0 µg/L

SECONDARY OUTCOMES:
Change in TBI | 6 months
  Total body iron (TBI)
Iron deficiency (TBI) | 6 months
  TBI <0.0 mg/kg
Iron deficiency (sTfr) | 6 months
  sTfr >8.3 μg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Villalpando, MD PhD, Principal Investigator — Instituto Nacional de Salud Publica (INSP)
Locations (1):
- Instituto Nacional de Salud Publica (INSP), Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finkelstein JL, Mehta S, Villalpando S, Mundo-Rosas V, Luna SV, Rahn M, Shamah-Levy T, Beebe SE, Haas JD. A Randomized Feeding Trial of Iron-Biofortified Beans on School Children in Mexico. Nutrients. 2019 Feb 12;11(2):381. doi: 10.3390/nu11020381. PMID 30759887